CLINICAL TRIAL: NCT04232852
Title: Probiotics and Systemic Inflammation in Patients With Metabolic Syndrome and High Cardiovascular Risk
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Arezina Kasti, Head of Clinical Nutrition Department, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ΕΒΔ427/12-06-2019
Record Dates: First submitted 2019-11-19; First posted 2020-01-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome; Cardiovascular Risk Factor
Keywords: metabolic syndrome; probiotics; cardiovascular risk factor
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Demographics, anthropometric measurements (weight, height, waist circumference, BMI) will be recorded, clinical data related to the patient's cardiovascular risk (MI with or without angioplasty, acute coronary syndrome with or without angioplasty). Systolic and diastolic pressure will be measured before and after the 12-week intervention.
  This group will receive a probiotic mix, which will contain strains of Streptococcus thermophilus, Saccharomyces cerevisiae, Lactobacillus acidophilus, L. rhamnosus L. helveticus, L. gasseri, L. plantarum, Bifidobacterium bifidum, Enterococcus faecium at a daily dose of 7 × 1010 CFU in the form of a capsule. During the intervention, participants will follow their eating habits as well as the physical activity of their personal routine, with the advice not to consume fermented dairy products.
  Interventions: Dietary Supplement: Probiotic mix
- Placebo supplement (Placebo Comparator): Demographics, anthropometric measurements (weight, height, waist circumference, BMI) will be recorded, clinical data related to the patient's cardiovascular risk (MI with or without angioplasty, acute coronary syndrome with or without angioplasty). Systolic and diastolic pressure will be measured before and after the 12-week intervention.
  Patients of this group will receive an identical capsule of maltodextrin (placebo). During the intervention, participants will follow their eating habits as well as the physical activity of their personal routine, with the advice not to consume fermented dairy products.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic mix — The probiotic mix will contain strains of Streptococcus thermophilus, Saccharomyces cerevisiae, Lactobacillus acidophilus, L. rhamnosus L. helveticus, L. gasseri, L. plantarum, Bifidobacterium bifidum, Enterococcus faecium at a daily dose of 7 × 1010 CFU in the form of a capsule.
  Arms: Probiotics
Dietary Supplement: Placebo — Patients in the placebo group will receive an identical capsule of maltodextrin.
  Arms: Placebo supplement

SUMMARY:
Metabolic Syndrome (MetS) and cardiovascular disease are associated with systemic inflammation (SI). Activation of the mechanisms of inflammation is triggered by the inflammatory cytokines. Τhe NLRP3 inflammasome is activated by microbial-derived low molecular weight (LMW) factors, short chain fatty acids (SCFAs), pathogen-associated molecular pattern molecules (PAMPs), damage-associated molecular pattern molecules (DAMPs), and monosodium urate crystals. Probiotics can regulate inflammation in two ways: 1) indirectly, by producing SCFAs as well as increasing synthesis of antimicrobial peptides and 2) directly, by binding innate immune system receptors Toll-like (TLR 2, 4, 9) and triggering important signaling pathways associated with activation of NLRs affecting the formation of inflammasome, thus the inflammatory response.

DETAILED DESCRIPTION:
Metabolic Syndrome (MetS) is associated with low-grade systemic inflammation (SI). Activation of the mechanisms of inflammation is triggered by the inflammatory cytokines produced in the adipose tissue. Among them, IL-1β interleukin plays a central role in cardiovascular disease. The active form of IL-1β results by the conversion of its inactive precursor after an infectious/inflammatory stimulus. The Nucleotide-binding Oligomerization Domain (NOD)-like Receptor containing Pyrin domain 3 (NLRP3 or cryopyrin) inflammasome is a multiprotein complex that activates caspase 1, leading to the processing and secretion of the pro-inflammatory cytokines interleukin-1β (IL-1β) via the NLRP3/caspase pathway. Τhe NLRP3 inflammasome is activated by microbial-derived Low Molecular Weight (LMW) factors, short chain fatty acids (SCFAs), Pathogen-associated molecular pattern molecules (PAMPs), Damage-associated molecular pattern molecules (DAMPs), and monosodium urate crystals.

It is a randomized, double-blind clinical trial in patients with MetS and cardiovascular disease. Patients will be randomized into two groups: A. those who will receive probiotic supplements and B. placebo-treated patients. Both groups will follow the usual clinical practice as far as drugs and diet concerned.

Τhe primary objective of this study is to investigate the effect of administration of the probiotic mix on IL-1β production by stimulated peripheral blood mononuclear cells (PBMCs) in patients at high cardiovascular risk with MetS at the end of the intervention. Secondly, to investigate the effect of probiotics on endothelial glycocalyx thickness, on hrCRP and on HbA1c levels, on the components of the MetS, on the gut microbiota at the end and 4 weeks after the completion of the intervention.

Time frame 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients≥50 years old, with diagnosed MetS and history of Myocardial Infarction (MI), angioplasty, acute coronary syndrome with or without angioplasty, after written consent.
* MetS syndrome defined by fulfilling at least 3 of the 5 following criteria: (NCEP-ATP-III) and "at high cardiovascular risk" as aforementioned.

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 40 (morbid obesity - difficult to manage, comorbidities)
* Probiotic intake three months prior to intervention
* Antibiotic intake three months prior to intervention
* Presence of inflammatory disease
* Inability to comply with study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
IL-1β production by stimulated peripheral blood mononuclear cells. | 12 weeks
  We will measure IL-1β concentrations in cell supernatants and consequently the NLRP3 inflammasome activation via the alteration in cytokine production in the presence of a different stimulants.
TNFα expression | 12 weeks
  Reverse Transcription Polymerase Chain Reaction (RT-PCR) will be used to quantify gene expression of tumor necrosis factor alpha (TNFα)
Caspase 1 (CASP1) expression | 12 weeks
  Reverse Transcription Polymerase Chain Reaction (RT-PCR) will be used to quantify CASΡ-1 as a key modulator of IL-1b bioactivity.

SECONDARY OUTCOMES:
Glycocalyx thikness. | 12 weeks
  The Perfused Boundary Region (PBR) of the hypoglossal vessels will be calculated using a high-resolution special lens using the Sideview DarkField (SDF) Imaging technique (Microscan, Glucockeck).
Change of biochemical exams related to MetS | 12 weeks
  Insulin resistance (IR) will be quantified using the HOMA-IR index (HOmeostatic Model Assessment, HOMA-IR index), calculated as the product of fasting plasma insulin. Blood lipids (Total Cholesterol, LDL-C, HDL-C, TRG) will be measured by enzymatic methods.
Alterations of hsCRP levels. | 12 weeks
  Hs-CRP will be measured by the Immunoturbidimetry method with a polyclonal antibody.
Alterations in gut microbiota | 12 weeks
  Stool specimen will be collected before and after intervention. Stool samples will be frozen (-80 ° C) immediately after collection, in order to study changes in the gut microbiota by the technique of deep sequencing at a second time.
Alterations of HbA1C | 12 weeks
  HbA1C will be measured by the HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Arezina Kasti, Principal Investigator — Attikon University General Hospital
Locations (1):
- Attikon University General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No